CLINICAL TRIAL: NCT02449135
Title: Nano Drug Interventional Therapy Using Digital Subtraction Angiography（DSA） for Pancreatic Carcinoma：Clinical Trial
Brief Title: Nano Drug Interventional Therapy Using Digital Subtraction Angiography（DSA） for Pancreatic Carcinoma
Status: No longer available | Type: Expanded Access
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: Nano drug pancreatic cancer
Record Dates: First submitted 2015-05-11; First posted 2015-05-20 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Nano drug
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Procedure: interventional therapy — Pancreatic cancer patients received drug interventional therapy using the digital subtraction angiography（DSA）.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nano drug interventional therapy using digital subtraction angiography（DSA） for pancreatic cancer. The nano drug is made by mixing Gemzar® with Compound Glycyrrhizin Injection.

DETAILED DESCRIPTION:
By enrolling patients with pancreatic cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of nano drug interventional therapy using digital subtraction angiography（DSA）for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80
2. Karnofsky performance status >60
3. Diagnosis of pancreatic cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive interventional therapy
6. Life expectancy: Greater than 3 months
7. Patients' routine blood test, liver function and kidney function have no obvious abnormalities
8. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except pancreatic cancer
2. History of coagulation disorders or anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Niu L, Chen J, Yao F, Zhou L, Zhang C, Wen W, Bi X, Hu Y, Piao X, Jiang F, Zeng J, Liu W, Li J, He L, Mu F, Zuo J, Xu K. Percutaneous cryoablation for stage IV lung cancer: a retrospective analysis. Cryobiology. 2013 Oct;67(2):151-5. doi: 10.1016/j.cryobiol.2013.06.005. Epub 2013 Jun 24. PMID 23806858
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Piao+xianghao